CLINICAL TRIAL: NCT02364713
Title: MC1365, A Randomized Phase II Trial of a Genetically Engineered NIS-Expressing Strain of Measles Virus Versus Investigator's Choice Chemotherapy for Patients With Platinum-Resistant Ovarian, Fallopian, or Peritoneal Cancer
Brief Title: MV-NIS or Investigator's Choice Chemotherapy in Treating Patients With Ovarian, Fallopian, or Peritoneal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1365; NCI-2015-00133 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1365 (Other: Mayo Clinic in Rochester); 14-000428 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Results first posted 2025-11-17 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-08

CONDITIONS: Fallopian Tube Carcinosarcoma; Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Fallopian Tube Undifferentiated Carcinoma; Ovarian Carcinosarcoma; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Adenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Adenocarcinoma; Ovarian Transitional Cell Carcinoma; Ovarian Undifferentiated Carcinoma; Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Ovarian Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma; Primary Peritoneal Carcinosarcoma; Primary Peritoneal Clear Cell Adenocarcinoma; Primary Peritoneal Endometrioid Adenocarcinoma; Primary Peritoneal Serous Adenocarcinoma; Primary Peritoneal Transitional Cell Carcinoma; Primary Peritoneal Undifferentiated Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Gemcitabine; Paclitaxel; Taxes; liposomal doxorubicin; Doxorubicin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (MV-NIS) (Experimental): Patients receive oncolytic measles virus encoding thyroidal sodium iodide symporter IP over 30 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Oncolytic Measles Virus Encoding Thyroidal Sodium Iodide Symporter; Other: Quality-of-Life Assessment
- Arm B (DOXIL, GEM, TOPA, TAXOL) (Active Comparator): Patients receive pegylated liposomal doxorubicin hydrochloride IV over 1 hour on day 1, or gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15, or topotecan hydrochloride IV over 30 minutes on days 1, 8, and 15, or paclitaxel IV over 1 hour on days 1, 8, and 15. Patients may also receive bevacizumab IV over 30-90 minutes on days 1 and 15 with pegylated liposomal doxorubicin hydrochloride, topotecan hydrochloride, or paclitaxel. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Other: Quality-of-Life Assessment; Drug: Topotecan Hydrochloride

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501
  Arms: Arm B (DOXIL, GEM, TOPA, TAXOL)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; FF 10832; FF-10832; FF10832; Gemcitabine HCI; Gemzar; LY-188011; LY188011
  Arms: Arm B (DOXIL, GEM, TOPA, TAXOL)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Oncolytic Measles Virus Encoding Thyroidal Sodium Iodide Symporter — Given IP
  Other Names: MV-NIS
  Arms: Arm A (MV-NIS)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm B (DOXIL, GEM, TOPA, TAXOL)
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; Dox-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
  Arms: Arm B (DOXIL, GEM, TOPA, TAXOL)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Hycamptamine; Hycamtin; SKF S-104864-A; Topotecan HCl; topotecan hydrochloride (oral)
  Arms: Arm B (DOXIL, GEM, TOPA, TAXOL)

SUMMARY:
This randomized phase II trial studies how well oncolytic measles virus encoding thyroidal sodium iodide symporter (MV-NIS) compared to investigator's choice chemotherapy works in treating patients with ovarian, fallopian, or peritoneal cancer. Measles virus, which has been changed in a certain way, may be able to kill tumor cells without damaging normal cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare clinical efficacy of Arm A (MV-NIS therapy) and Arm B (standard cytotoxic chemotherapy), as measured by overall survival (OS).

SECONDARY OBJECTIVES:

I. Compare progression-free survival (PFS), overall survival at 12 months (OS12), progression-free survival at six months (PFS6), and objective response rate (ORR) between MV-NIS therapy and standard chemotherapy.

II. Assess safety and tolerability of MV-NIS, and compare with standard chemotherapy.

III. Compare quality of life as assessed by Functional Assessment of Cancer Therapy-Ovarian (FACT-O) between MV-NIS and standard chemotherapy.

TRANSLATIONAL OBJECTIVES:

I. Assess the time course of viral gene expression and virus elimination and biodistribution of virally infected cells at various time points after infection with MV-NIS using single-photon emission computerized tomography (SPECT)/computed tomography (CT) imaging within the MV-NIS treatment arm.

II. Assess viremia, viral replication, and viral shedding/persistence following intraperitoneal administration within the NV-NIS treatment arm.

III. Measure humoral and cellular immune responses to MV-NIS within the NV-NIS treatment arm.

IV. Measure changes in anti-ovarian cancer (OC) immune responses in both treatment arms.

V. Perform transcriptomic analysis on tumor biopsy specimens to determine a gene expression profile predictive of therapeutic response to MV-NIS.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive oncolytic measles virus encoding thyroidal sodium iodide symporter intraperitoneally (IP) over 30 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive pegylated liposomal doxorubicin hydrochloride intravenously (IV) over 1 hour on day 1, or gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15, or topotecan hydrochloride IV over 30 minutes on days 1, 8, and 15, or paclitaxel IV over 1 hour on days 1, 8, and 15. Patients may also receive bevacizumab IV over 30-90 minutes on days 1 and 15 with pegylated liposomal doxorubicin hydrochloride, topotecan hydrochloride, or paclitaxel. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months until disease progression and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION INCLUSION CRITERIA:
* Ability to understand and the willingness to sign a written informed consent document
* The effects of the candidate chemoprevention agents on the developing human fetus remain incompletely defined; however, study participants will be women who have gone through a bi-lateral oophorectomy procedure
* Willingness to be evaluated for surgical placement of an intraperitoneal port and undergo biopsy if feasible for a research sample
* REGISTRATION/RANDOMIZATION INCLUSION CRITERIA:
* Recurrent, persistent, or progressive epithelial ovarian, fallopian tube, or primary peritoneal cancer after treatment with bilateral oophorectomy and either cisplatin or carboplatin and either paclitaxel, albumin-bound paclitaxel, or docetaxel; histologic confirmation of the primary tumor is required; eligible histologies include serous, endometrioid, clear cell, mucinous, transitional cell, undifferentiated, or mixed carcinoma
* Platinum-resistant or platinum-refractory disease, defined as either 1) less than a complete response to the most recent carboplatin- or cisplatin-containing chemotherapy regimen, 2) serum cancer antigen (CA)-125 >= 2 x upper limit of normal (ULN) within 180 days of last dose of carboplatin- or cisplatin-containing chemotherapy, confirmed by a second CA-125 (the second CA-125 does not have to be within 180 days of chemotherapy), or 3) CT or positron emission tomography (PET)/CT evidence of cancer recurrence within 180 days of last dose of carboplatin- or cisplatin-containing chemotherapy
* Absolute neutrophil count (ANC) >= 1500/uL (obtained =< 7 days prior to registration)
* Platelet (PLT) >= 100,000/uL (obtained =< 7 days prior to registration)
* Total bilirubin =< ULN (obtained =< 7 days prior to registration)
* Aspartate aminotransferase (AST) =< 2 x ULN (obtained =< 7 days prior to registration)
* Creatinine =< 1.5 x ULN (obtained =< 7 days prior to registration)
* Hemoglobin (Hgb) >= 9.0 g/dL (obtained =< 7 days prior to registration)
* Willingness to return to Mayo Clinic Rochester or another participating institution for follow-up; patients who are randomized to Arm B (cytotoxic chemotherapy) may receive chemotherapy at any oncology clinic able to provide the protocol-directed therapy and willing to send laboratory data to the participating institution; however, patients must be willing to return to the participating institution every two months for evaluation; patients who are randomized to Arm A must be willing to receive all treatment and follow-up at a participating institution
* Life expectancy >= 12 weeks
* Willingness to provide all biologic specimens as required by the protocol
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria, or evaluable disease by CA-125; (NOTE: CA-125-evaluable disease is defined as serum CA-125 >= 2 x ULN that is determined by the treating clinician to be due to recurrent ovarian, fallopian tube, or primary peritoneal cancer)
* Normal cardiac function, as determined by left ventricular ejection fraction (LVEF) >= institutional lower limit of normal on echocardiogram or multi-gated acquisition scan (MUGA) =< 1 month prior to registration
* If liposomal doxorubicin hydrochloride (DOXIL) is selected as the investigator's choice chemotherapy:

  * Lifetime exposure to doxorubicin =< 240 mg/m^2 (or equivalent biologic dose if prior exposure to a different anthracycline)
* Candidate for surgical placement of an intraperitoneal port, as determined by a gynecologic oncology surgeon
* Must have anti-measles immunity as demonstrated by serum immunoglobulin (Ig)G anti-measles antibody levels of >= 1.1 EU/ml as determined by BioPlex Measles IgG multiplex flow immunoassay

Exclusion Criteria:

* REGISTRATION/RANDOMIZATION EXCLUSION CRITERIA:
* Epithelial tumors of low malignant potential, stromal tumors, and germ cell tumors of the ovary
* Evidence of measurable disease (per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST 1.1]) outside of the peritoneal cavity (ex: mediastinal lymphadenopathy, parenchymal liver metastasis, or symptomatic pleural effusion proven or suspected to be due to cancer)

  * Note: Asymptomatic pleural effusion with or without minimal pleural involvement as long as there is no measurable disease outside the peritoneum/retroperitoneum is allowed
* Bulky metastases, defined as any tumor nodule or lymph nodes > 5 cm in greatest dimension on axial images on pre-treatment CT, PET/CT, or magnetic resonance imaging (MRI)

  * Note: patients with bulky (> 5 cm) disease for whom gross total cytoreduction is deemed feasible by a surgeon (with confirmation by a second surgeon after radiologic review) are eligible for participation in the context of cytoreductive surgery
* Resistant to all of the following: DOXIL, gemcitabine hydrochloride (GEM), topotecan hydrochloride (TOPA), and weekly paclitaxel (TAXOL); (NOTE: resistance is defined as either 1) less than a complete response to any chemotherapy regimen containing the agent in question [consider weekly TAXOL as a separate agent from every-three-week TAXOL], 2) serum CA-125 >= 2 x ULN within 180 days of last dose of chemotherapy containing the agent in question, confirmed by a second CA-125 [the second CA-125 does not have to be within 180 days of chemotherapy], or 3) CT or PET/CT evidence of cancer recurrence/progression within 180 days of last dose of chemotherapy containing the agent in question; [for example, if a patient previously received carboplatin and GEM, had a complete response, and had initial evidence of relapse > 180 days after the last dose of GEM, that patient would not be considered resistant to GEM])
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 3 or 4
* History of other malignancy =< 5 years prior to registration except for non-melanoma skin cancer, carcinoma in situ of the cervix, and ductal carcinoma in situ (DCIS)
* Active infection =< 7 days prior to study entry
* Any of the following prior therapies:

  * Chemotherapy =< 3 weeks prior to study entry
  * Immunotherapy =< 4 weeks prior to study entry
  * Biologic therapy =< 4 weeks prior to study entry
  * Extensive abdominal surgery if it includes enterotomy(ies) =< 3 weeks prior to study entry; (NOTE: this criterion does not apply to placement of the peritoneal Port-A-Cath or lysis of adhesions at the time of study entry)
  * Any viral or gene therapy prior to study entry
* Failure to recover to =< grade 1 from acute, reversible effects of prior chemotherapy, excluding alopecia regardless of interval since last treatment; (NOTE: patients with residual peripheral neuropathy are allowed)
* New York Heart Association classification III or IV congestive heart failure, known symptomatic coronary artery disease, symptoms of coronary artery disease on systems review, or known cardiac arrhythmias (atrial fibrillation or supraventricular tachycardia [SVT])
* Other cardiac or pulmonary disease that, at the investigator's discretion, can impair treatment safety
* Central nervous system (CNS) metastases or seizure disorder
* Human immunodeficiency virus (HIV)-positive test result, or history of other immunodeficiency
* History of organ transplantation
* History of chronic hepatitis B or C
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Any concurrent medications which could interfere with the trial
* History of tuberculosis or history of purified protein derivative (PPD) positivity
* Treatment with oral/systemic corticosteroids, with the exception of topical or inhaled steroids or steroids given for the purpose of adrenal replacement given at physiologic doses
* Exposure to household contacts =< 15 months old or household contact with known immunodeficiency
* Allergy to measles vaccine or history of severe reaction to prior measles vaccination
* Allergy to iodine; (NOTE: this does not include reactions to intravenous contrast materials)
* Any other pathology or condition which the principal investigator may deem to negatively impact treatment safety
* On anticoagulation and unable to discontinue temporarily for up to 7 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-03-13 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (MV-NIS): Patients receive oncolytic measles virus encoding thyroidal sodium iodide symporter IP over 30 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.>
  > Laboratory Biomarker Analysis: Correlative studies>
  > Oncolytic Measles Virus Encoding Thyroidal Sodium Iodide Symporter: Given IP>
  > Quality-of-Life Assessment: Ancillary studies
- Arm B (DOXIL, GEM, TOPA, TAXOL): Patients receive pegylated liposomal doxorubicin hydrochloride IV over 1 hour on day 1, or gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15, or topotecan hydrochloride IV over 30 minutes on days 1, 8, and 15, or paclitaxel IV over 1 hour on days 1, 8, and 15. Patients may also receive bevacizumab IV over 30-90 minutes on days 1 and 15 with pegylated liposomal doxorubicin hydrochloride, topotecan hydrochloride, or paclitaxel. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.>
  > Bevacizumab: Given IV>
  > Gemcitabine Hydrochloride: Given IV>
  > Laboratory Biomarker Analysis: Correlative studies>
  > Paclitaxel: Given IV>
  > Pegylated Liposomal Doxorubicin Hydrochloride: Given IV>
  > Quality-of-Life Assessment: Ancillary studies>
  > Topotecan Hydrochloride: Given IV
Period: Overall Study
Arm/Group | Arm A (MV-NIS) | Arm B (DOXIL, GEM, TOPA, TAXOL)
Started | 10 | 7
Completed | 8 | 5
Not Completed | 2 | 2
Not completed — Ineligible | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (MV-NIS) | Arm B (DOXIL, GEM, TOPA, TAXOL) | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Continuous [Median (Full Range); unit: years] | 68 [57 to 83] | 64 [39 to 78] | 67 [39 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 6 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Defined as the time from registration/randomization to death due to all causes. Will be a comparison of the oncolytic measles virus encoding thyroidal sodium iodide symporter versus investigator's choice chemotherapy using a one-sided log-rank test.
Time Frame: 5 years
Population: All eligible and treated patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (MV-NIS) | Arm B (DOXIL, GEM, TOPA, TAXOL)
Number analyzed (Participants) | 8 | 5
Months | 11.2 [3.5 to NA] — Too few events to calculate the upper limit | 14.2 [10.6 to NA] — Too few events to calculate the upper limit

2. Secondary Outcome: Progression-free Survival
Description: Defined as the time from start of study therapy to the date of first observation of disease progression or death due to any cause (whichever comes first). The distribution of progression-free survival for both arms of the study will be estimated using the Kaplan-Meier method.
Time Frame: 11 months
Population: All eligible and treated patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (MV-NIS) | Arm B (DOXIL, GEM, TOPA, TAXOL)
Number analyzed (Participants) | 8 | 5
Months | 1.8 [1.7 to NA] — Too few events to calculate the upper limit | 4.1 [1.8 to NA] — Too few events to calculate the upper limit

3. Secondary Outcome: Overall Survival
Description: Defined as the time from registration/randomization to death due to all causes. Overall survival at 12 months distributions both arms of the study will be estimated using the Kaplan-Meier method and be compared using a one-sided logrank test.
Time Frame: 12 months
Population: All eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (MV-NIS) | Arm B (DOXIL, GEM, TOPA, TAXOL)
Number analyzed (Participants) | 8 | 5
Participants | 4 | 2

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival at 6 months distributions both arms of the study will be estimated using the Kaplan-Meier method.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (MV-NIS) | Arm B (DOXIL, GEM, TOPA, TAXOL)
Number analyzed (Participants) | 8 | 5
Participants | 5 | 4

5. Secondary Outcome: Objective Response Rate
Description: Objective response rate is defined to be a complete response or partial response noted as the objective status on 2 consecutive evaluations at least 4 weeks apart
Time Frame: 11 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (MV-NIS) | Arm B (DOXIL, GEM, TOPA, TAXOL)
Number analyzed (Participants) | 8 | 5
Participants | 0 | 0

6. Secondary Outcome: Incidence of Adverse Events Per Common Terminology Criteria for Adverse Events Version 4.0
Description: Safety and tolerability of the oncolytic measles virus encoding thyroidal sodium iodide symporter as compared to standard therapy will be evaluated using all patients who have received any study treatment as well as summarizing those who have been included in the efficacy analyses. The overall adverse event rates for grade 3 or higher adverse events will be compared between arms.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (MV-NIS) | Arm B (DOXIL, GEM, TOPA, TAXOL)
Number analyzed (Participants) | 8 | 5
Participants | 3 | 2

7. Secondary Outcome: Quality of Life as Measured by the Functional Assessment of Cancer Therapy-Ovarian Questionnaire
Description: Quality of life as measured by the Functional Assessment of Cancer Therapy-Ovarian (FACT-O) questionnaire will be compared between treatment arms. The assessment will be scored according to the assessment scoring algorithm at each collection time. Scores at end of each cycle will be compared using Wilcoxon procedures. The FACT-O consist of 39 questions, each answered on a 5-point Likert scale ranging from 0 (Not at all) to 4 (Very much). Possible total scores range from 0-156, with higher scores indicating better quality of life. We will calculate the mean change from the start to the end of the study of patient total FACT-O point sum by arm.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: change in score
Arm/Group | Arm A (MV-NIS) | Arm B (DOXIL, GEM, TOPA, TAXOL)
Number analyzed (Participants) | 6 | 3
change in score | 5.2 (14.6) | -12.6 (12.1)

8. Other Pre Specified Outcome: Time Course of Viral Gene Expression and Virus Elimination and Biodistribution of Virally Infected Cells Using Single-photon Emission Computerized Tomography/Computed Tomography Imaging
Description: Descriptive statistics and simple scatter plots will form the basis of presentation of these data. Correlations between these laboratory values and other outcome measures will be carried out by standard parametric and nonparametric correlation procedures (Pearson's and Spearman's coefficients).
Time Frame: Up to course 2
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Viremia, Viral Replication, and Viral Shedding/Persistence Following Intraperitoneal Administration Within the Oncolytic Measles Virus Encoding Thyroidal Sodium Iodide Symporter Treatment Arm
Description: as for outcome 8
Time Frame: Up to 5 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Humoral and Cellular Immune Responses to Oncolytic Measles Virus Encoding Thyroidal Sodium Iodide Symporter
Description: as for outcome 8
Time Frame: Up to 5 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Changes in Anti-ovarian Cancer Immune Responses in Both Treatment Arms
Description: as for outcome 8
Time Frame: Baseline to up to 5 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Gene Expression Profile Predictive of Therapeutic Response to Oncolytic Measles Virus Encoding Thyroidal Sodium Iodide Symporter
Description: as for outcome 8
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were followed for 12 months and mortality was followed for 5 years
Description: All accrued patients are included in mortality reporting. All treated patients are included in the adverse events, this includes a patient that's been deemed ineligible.
Arm/Group | Arm A (MV-NIS) | Arm B (DOXIL, GEM, TOPA, TAXOL)
All-Cause Mortality (participants affected / at risk) | 8/10 | 5/7
Serious Adverse Events (participants affected / at risk) | 6/9 | 2/5
Other Adverse Events (participants affected / at risk) | 8/9 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (MV-NIS) (N=9) | Arm B (DOXIL, GEM, TOPA, TAXOL) (N=5)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (MV-NIS) (N=9) | Arm B (DOXIL, GEM, TOPA, TAXOL) (N=5)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (6) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (2)
Vomiting (Gastrointestinal disorders) | 5 (7) | 1 (2)
Chills (General disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 3 (6) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (5)
Platelet count decreased (Investigations) | 1 (5) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 3 (9)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (2)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT02364713/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/13/NCT02364713/ICF_001.pdf